CLINICAL TRIAL: NCT06867822
Title: A Phase I/Ib Trial of ProAgio, an Anti-avb3 Integrin Cytotoxin, in Combination With 5-fluorouracil , Irinotecan and Bevacizumab for Advanced/Metastatic Colorectal Cancer (ProAgio in CRC)
Brief Title: Trial of ProAgio in Advanced/Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: The V Foundation (Other)
Responsible Party: Principal Investigator, Midhun Malla, MD, Associate Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300014432 (UAB2479); T2024-020 (Other Grant/Funding Number: V Foundation)
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Advanced Colorectal Cancer; Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — IFL protocol; Fluorouracil; Leucovorin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase I: dose escalation ProAgio + FOLFIRI + bevacizumab dose levels tested for RP2D (Experimental): Dose level ProAgio mg/Kg FOLFIRI + bevacizumab
  1. MTD-2 (6.4*) FOLFIRI + bevacizumab
  2. MTD-1 (10.7) FOLFIRI + bevacizumab
  3. MTD (12.5) FOLFIRI + bevacizumab
  4. MTD+1 (16*) FOLFIRI + bevacizumab
  ProAgio will be administered via IV over 60 minutes on Day 1, 8, 15, and 21 every 4-week cycle.
  Bevacizumab 5 mg/kg, Irinotecan 180 mg/m2, 5-Flurouracil infusion 2400 mg/m2 will be administered via IV on Day 1, and 15 every 4-week cycle.
  The study will use an Accelerated titration BOIN design in Phase I to determine the recommended RP2D of ProAgio with FOLFIRI + bevacizumab. The trial will estimate the RP2D of ProAgio when combined with FOLFIRI + bevacizumab, starting from 2 dose levels lower than the estimated RP2D of ProAgio alone. Accelerated titration BOIN design will enroll patients with the 4 combination dose levels listed above, maximum of 15 subjects.
  Interventions: Drug: ProAgio; Drug: FOLFIRI; Drug: Bevacizumab
- Phase Ib: dose expansion ProAgio + FOLFIRI + bevacizumab (Experimental): Once the MTD and RP2D of ProAgio with FOLFIRI have been identified, an expansion cohort of 12 subjects with advanced/metastatic CRC will begin. The purpose of the expansion cohort is to confirm the safety of the regimen and provide preliminary data on the activity of ProAgio + FOLFIRI + bevacizumab.
  Interventions: Drug: ProAgio; Drug: FOLFIRI; Drug: Bevacizumab

INTERVENTIONS:
Drug: ProAgio — ProAgio is a pegylated protein with a single pegylated site. The 12,131 Dalton protein is produced in E. coli and is composed of 105 amino acids with no disulfide bonds. The structure of the polyethylene glycol moiety is Methoxy PEG maleimide 30000.
  Other Names: ACT50
Drug: FOLFIRI — FOLFIRI is a combination of three drugs: (leucovorian, fluorouracil, and irinotecan) used to treat advanced metastatic colorectal cancer. FOLFIRI is commercially available will be administered using standard dosing regimen as per institutional guidelines.
  Other Names: Irinatecan; 5-fluorouracil; folinic acid (leucovorin)
Drug: Bevacizumab — Bevacizumab is a recombinant humanized monoclonal antibody that blocks angiogenesis by inhibiting vascular endothelial growth factor A (VEGF-A). Bevacizumab is commercially available and will be administered using standard dosing regimen as per institutional guidelines.
  Other Names: Avastin

SUMMARY:
This is an open-label Phase I/Ib dose-escalation, dose-expansion clinical trial of the safety, pharmacokinetics and clinical activity of ProAgio combined with 5-fluorouracil, irinotecan (FOLFIRI) and bevacizumab for untreated advanced/metastatic CRC. The study will use an Accelerated titration BOIN design in Phase I to determine the recommended RP2D of ProAgio with FOLFIRI + bevacizumab. The trial will estimate the RP2D of ProAgio when combined with FOLFIRI + bevacizumab, starting from 2 dose levels lower than the estimated RP2D of ProAgio alone. Accelerated titration BOIN design will enroll patients with the 4 combination dose levels.

Subjects will be selected based on following criteria: previously untreated advanced/metastatic CRC, ECOG performance status (0-1), and adequate organ functions. Subjects with recent surgeries, history of recent thromboembolic events or significant cardiovascular disease will be excluded.

Once the MTD and RP2D of ProAgio with FOLFIRI have been identified, an expansion cohort of 12 subjects with advanced/metastatic CRC will begin. The purpose of the expansion cohort is to confirm the safety of the regimen and provide preliminary data on the activity of ProAgio + FOLFIRI + bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥18 years of age at the time of consent.
2. Histologic or cytologic diagnosis of colorectal adenocarcinoma (CRC)
3. Patients with advanced or metastatic CRC
4. Performance status, ECOG: 0, 1
5. For dose escalation phase: patients with CRC where FOLFIRI+ bevacizumab is considered appropriate standard therapy (previously treated with FOLFOX based regimen in advanced/metastatic CRC is allowed). For dose expansion phase: patients must not have received 5FU-based therapy previously for metastatic disease. Patients who received FOLFOX/CAPOX regimens in the neoadjuvant/adjuvant setting are allowed if recurrence free survival is at least 1 year or longer since completion of adjuvant therapy.
6. Presence of a metastatic lesion that can be safely biopsied for correlative assays (Only for FOUR patients enrolling on the dose expansion phase).
7. Patient must meet the following laboratory values at the screening visit:

   * Absolute Neutrophil Count ≥1.5 x 109/L
   * Platelets ≥100 x 109/L
   * Hemoglobin (Hgb) ≥9 g/dL
   * Creatinine Clearance ≥60 mL/min using Cockcroft-Gault formula
   * Total bilirubin ≤1.5 x ULN
   * Aspartate transaminase (AST) ≤2.5 x ULN, except for subjects with liver metastasis, who may only be included if AST ≤5.0 x ULN
   * Alanine transaminase (ALT) ≤2.5 x ULN, except for subjects with liver metastasis, who may only be included if ALT ≤5.0 x ULN
   * Urine dipstick reading for proteinuria < 2+. Participants having ≥ 2+ proteinuria on urine dipstick testing at baseline will undergo a 24-hour urine collection for quantitative assessment of proteinuria and must demonstrate < 1 g of protein in 24 hours. Participants with urine protein ≥ 1 g per 24 hours will be ineligible
8. Blood pressure <=160/100 mm Hg
9. Presence of measurable disease by RECIST 1.1 criteria within 28 days prior to the first dose of study treatment.
10. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status 0- 1 (Appendix A-Performance Status Criteria).
11. Normal ECG defined as the following: QTcF at screening <450 ms (male subjects), <460 ms (female subjects)
12. Before enrollment, a woman must be either:

    1. Not of childbearing potential: postmenopausal (>45 years of age with amenorrhea for at least 12 months or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level >40 IU/mL); permanently sterilized (eg, tubal occlusion, hysterectomy, bilateral salpingectomy); or otherwise be incapable of pregnancy.
    2. Of childbearing potential and practicing (during the study and for 6 months after receiving the last dose of study agent for women and 3 months after receiving the last dose of study agent for men)) a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies: e.g., established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device (IUD) or intrauterine system (IUS); barrier methods; true abstinence (when this is in line with the preferred and usual lifestyle of the subject).
    3. Note: If the childbearing potential changes after start of the study (eg, woman who is not heterosexually active becomes active) a woman must begin a highly effective method of birth control, as described above.
13. A woman of childbearing potential must have a negative serum (β-human chorionic gonadotropin [β-hCG]) or urine pregnancy test at screening.
14. During the study and for 6 months after receiving the last dose of study agent, a woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction.
15. A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control e.g., either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 3 months after receiving the last dose of study drug.
16. Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written informed consent and privacy language as per HIPAA must be obtained from the subject or legally authorized representative (if applicable) prior to any study- related procedures
17. Sign an informed consent document indicating that they understand the purpose of and procedures required for the study, are willing to participate in the study, and are willing and able to adhere to the prohibitions and restrictions specified in this protocol. Informed consent must be obtained before performing any study specific procedures.
18. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study
19. Subject agrees not to participate in another interventional study while receiving study drug in present study

Exclusion Criteria:

1. Prior exposure to FOLFIRI chemotherapy
2. Clinically significant peripheral neuropathy (>=Grade 3 per CTCAE 5.0)
3. Any untreated central nervous system (CNS) lesion. However, subjects are eligible if: a) all known CNS lesions have been treated with radiotherapy or surgery and b) patient remained without evidence of CNS disease progression ≥4 weeks after treatment.
4. Allogenic bone marrow or solid organ transplant
5. Known history or current interstitial lung disease or non-infectious pneumonitis
6. Prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen, per treating physician discretion.
7. Known additional malignancy that is progressing or requires active treatment, with the exception of patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or antitumor assessment of the investigational regimen.
8. Subject has known dihydropyrimidine dehydrogenase (DPD) deficiency. (NOTE: DPD testing is not mandatory as part of the trial and can be performed at the discretion of treating provider per local requirements)
9. Subject has known immediate or delayed hypersensitivity, intolerance or contraindication to any component of study treatment
10. Infection with human immunodeficiency virus (HIV)-1 or HIV-2. (Exception:

    Participants with well-controlled HIV [ie, CD4 > 350/mm3 and undetectable viral load] are eligible.)
11. Active hepatitis, including the following:

    1. Acute or chronic hepatitis B (Exception: Participants who are hepatitis B surface antigen [HbsAg] positive are eligible if they have hepatitis B virus (HBV) DNA less than 500 IU/mL or 2,500 copies/mL). Note: Participants with detectable HbsAg or detectable HBV DNA should be managed per institutional or local standards. Participants beginning antiviral agents at screening should be treated for > 2 weeks prior to expected date of C1D1.
    2. Infection with hepatitis C (Exceptions: [i] Participants who have no history of curative viral treatment and are documented to be viral load negative are eligible; [ii] Participants who have completed curative viral therapy ≥ 12 weeks prior to expected date of C1D1, and viral load is negative are eligible.)
12. Severe chronic or active infections requiring systemic parenteral antibacterial, antifungal or antiviral therapy; or any other potentially life-threatening viral or bacterial infection (participants on oral antibiotics must complete the planned course of treatment prior to expected date of C1D1).
13. Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 14 days or 5 half-lives before enrollment or is currently enrolled in the treatment stage of an investigational study.
14. A woman who is pregnant or breast-feeding, or a woman who is planning to become pregnant or a man who plans to father a child while enrolled in this study or within 150 days after the last dose of study agent.
15. Subject has had a major surgical procedure ≤ 28 days prior to randomization. Subject without complete recovery from a major surgical procedure ≤ 14 days prior to randomization
16. Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
17. Subject has psychiatric illness or social situations such as incarceration that would preclude study compliance, per investigator judgment
18. Patients with a history of perforation, fistula, life-threatening gastrointestinal bleeding, proteinuria (>1 gm/24 hours), wound healing issues
19. Subject has significant cardiovascular disease, including any of the following:

    1. Congestive heart failure (defined as New York Heart Association [NYHA] Class III or IV), myocardial infarction, unstable angina, coronary angioplasty, coronary stenting, coronary artery bypass graft, cerebrovascular accident (CVA), or hypertensive crisis within 6 months prior to randomization;
    2. History of clinically significant ventricular arrhythmias (i.e., sustained ventricular tachycardia, ventricular fibrillation, or Torsades de Pointes);
    3. History or family history of congenital long QT syndrome
    4. Cardiac arrhythmias requiring anti-arrhythmic medications (Subjects with rate controlled atrial fibrillation for > 1 month prior to randomization are eligible.)
    5. Deep venous thrombosis/pulmonary embolism (within last 6 months) unless adequately treated with therapeutic anticoagulation.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change in NCI CTCAE scale version 5.0 | Baseline, up to 18 months
  National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE.

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics of ProAgio | Baseline, up to 10 months
  Assessed by measurement of serum levels of ProAgio over time following IV infusion.
Assessment of anti-tumor activity by measuring objective response rate (ORR) | up to 12 weeks
  The proportion of participants with partial response or complete response. RECIST 1.1 will be used to assess ORR.
Progression free survival (PFS) - duration of time from start of treatment to time of progression or death, whichever occurs first. | up to 18 months
  Determined from date of 1st dose of study drug to disease progression and/or death from any cause.
Overall survival (OS) - the length of time from start of treatment until death from any cause. | up to 18 months
  Determined from date of 1st dose of study drug to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States